CLINICAL TRIAL: NCT02141841
Title: Effect of Age on the Median Effective Concentration(EC50) for Motor Block With Spinal Plain Bupivacaine
Status: Withdrawn | Type: Observational
Why Stopped: because the study is very complicated and cannot be performed in the practice
Sponsor: China Three Gorges University, Yichang, China (Other)
Responsible Party: Principal Investigator, Mingquan Chen, China Three Gorges University, Yichang, China, China Three Gorges University, Yichang, China
Other Study IDs: China Three Gorges University
Record Dates: First submitted 2014-05-13; First posted 2014-05-20 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Mononeuropathy of the Median Nerve, Mild
Keywords: intrathecal;; bupivacaine;; concentration;
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study was performed in 131 adult patients undergoing transurethral, urological or lower limb surgery under combined spinal and epidural anesthesia. Patients were stratified according to age: 20-30, 31-40, 41-50, 51-60, 61-70, and 71-80 years. The spinal component of the anesthetic was established by bolus administration of up-and-down doses of 0.75% plain bupivacaine, determined by Dixon's method. The degree of motor block after intrathecal administration of each concentration was evaluated by the modified Bromage and Hip motor function score. The EC50 were estimated from the up-and-down sequences using the method of Dixon and Massey and logistic regression. Other endpoints were included on the basis of sensory block level, duration of motor blockade, hypotension, and vasopressor requirements.

ELIGIBILITY:
Inclusion Criteria:

- ASA physical status I-II adult patients who were undergoing transurethral, urological or lower limb surgery, primarily under the spinal component of established combined epidural-spinal anesthesia, with the epidural component to be used if there was a need for intra-operative analgesic supplementation or for postoperative analgesia.

Exclusion Criteria:

* Patients with diabetes, obesity, neuromuscular diseases, bleeding diathesis, hypersensitivity to amide local anesthetics, lumbar vertebrae abnormality, chronic back pain, or who were pregnant were excluded from this study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was performed in 131 adult patients undergoing transurethral, urological or lower limb surgery under combined spinal and epidural anesthesia.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
the median effect concentration of bupivacaine | The endpoint was determined according to the degree of motor power in any lower limb (according to the modified Bromage scale and the Hip motor function scale) within 5 minutes after intrathecal administration of the tested bupivacaine concentration
  The endpoint was determined according to the degree of motor power in any lower limb (according to the modified Bromage scale and the Hip motor function scale) within 5 minutes after intrathecal administration of the tested bupivacaine concentration
sensory block level | 20 minutes
  the sensory level was assessed by the pinprick or ice at interval 5 minutes and 2 0minutes after injection of spinal bupivacaine.

CONTACTS AND LOCATIONS:
Locations (1):
- China Three Gorges University, Yichang, Hubei, China

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/24651241